CLINICAL TRIAL: NCT07181031
Title: Comparative Effects of High-Intensity Interval and Functional Training on Performance Outcomes in Adolescent Female Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duvenciler Anadolu Lİsesi (Other)
Responsible Party: Principal Investigator, Omer Faruk Bilici, Principal Investigator, Duvenciler Anadolu Lİsesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09.2021.06
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Youth Volleyball; Sports Performance; Neuromuscular Function; Aerobic Capacity; Explosive Strength; Agility; Motor Skill Development
Keywords: High-Intensity Interval Training; High-Intensity Functional Training; Explosive Strength; Strength Training; Sports Performance
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Thirty-two adolescent female volleyball players were randomly assigned into three parallel groups: high-intensity interval training (HIIT, n=10), high-intensity functional training (HIFT, n=11), or control (n=11). The intervention period lasted 12 weeks, with two supervised training sessions per week in addition to routine volleyball practices. Pre- and post-tests were conducted to evaluate physical, physiological, and volleyball-specific performance outcomes.
Masking Description: No masking was applied; both participants and investigators were aware of group assignments (HIIT, HIFT, or control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-Intensity Interval Training (HIIT) (Experimental): Participants in the HIIT group engaged in a 12-week resistance-based high intensity interval training program, designed to target both aerobic and anaerobic energy systems. Training sessions were conducted twice per week in addition to the athletes' regular volleyball practice schedule. Each session commenced with a standardized 10-minute warm-up involving low-intensity jogging and dynamic stretching, and concluded with a 5-minute cool-down of light jogging and static stretching to promote recovery. The main training component consisted of short, repeated high intensity bouts (30 s) of multi-modal exercises-including sprint drills, plyometric movements, functional bodyweight resistance exercises, multi-joint strength movements, agility drills, and aerobic conditioning-performed at 85-95% of maximal heart rate (HRmax) [28,13]. Each bout was followed by 30 s of active recovery (e.g., walking or light movement).
  Interventions: Behavioral: High-Intensity Interval Training (HIIT)
- High-Intensity Functional Training (HIFT) (Experimental): Participants completed a 12-week high intensity functional training program aimed at developing aerobic capacity, anaerobic power, muscular strength, and agility. Training sessions were performed twice weekly in addition to regular volleyball practices. Each training session followed a standardized structure, beginning with a 10-minute warm-up of light jogging and dynamic mobility exercises, followed by a main training phase consisting of circuit-style functional workouts that combined sprint drills, plyometric exercises, bodyweight resistance movements, multi-joint strength exercises, agility drills, and aerobic activities; each exercise was performed for 30 seconds at maximal effort with no fixed rest between exercises (≤10 seconds transition allowed), and participants completed 4-6 sets per session with 1-2 minutes of rest between sets, while emphasizing maximal movement speed and explosive execution of all repetitions, and concluding with a 5-minute cool-down of low-intensity jogg
  Interventions: Behavioral: High-Intensity Functional Training (HIFT)
- Control (Routine Volleyball Training) (No Intervention): articipants continued their standard volleyball training program (3-4 sessions per week). To balance training exposure, they also completed the same number of additional supervised sessions as the intervention groups, consisting of regular volleyball practice only, without HIIT or HIFT conditioning.

INTERVENTIONS:
Behavioral: High-Intensity Interval Training (HIIT) — Participants in the HIIT group engaged in a 12-week resistance-based high intensity interval training program, designed to target both aerobic and anaerobic energy systems. Training sessions were conducted twice per week in addition to the athletes' regular volleyball practice schedule. Each session commenced with a standardized 10-minute warm-up involving low-intensity jogging and dynamic stretching, and concluded with a 5-minute cool-down of light jogging and static stretching to promote recovery. The main training component consisted of short, repeated high intensity bouts (30 s) of multi-modal exercises-including sprint drills, plyometric movements, functional bodyweight resistance exercises, multi-joint strength movements, agility drills, and aerobic conditioning-performed at 85-95% of maximal heart rate (HRmax) [28,13]. Each bout was followed by 30 s of active recovery (e.g., walking or light movement).
  Other Names: Resistance-based HIIT
  Arms: High-Intensity Interval Training (HIIT)
Behavioral: High-Intensity Functional Training (HIFT) — Participants completed a 12-week high intensity functional training program aimed at developing aerobic capacity, anaerobic power, muscular strength, and agility. Training sessions were performed twice weekly in addition to regular volleyball practices. Each training session followed a standardized structure, beginning with a 10-minute warm-up of light jogging and dynamic mobility exercises, followed by a main training phase consisting of circuit-style functional workouts that combined sprint drills, plyometric exercises, bodyweight resistance movements, multi-joint strength exercises, agility drills, and aerobic activities; each exercise was performed for 30 seconds at maximal effort with no fixed rest between exercises (≤10 seconds transition allowed), and participants completed 4-6 sets per session with 1-2 minutes of rest between sets, while emphasizing maximal movement speed and explosive execution of all repetitions, and concluding with a 5-minute cool-down of low-intensity joggi
  Other Names: High Intensity Functional Circuit Training
  Arms: High-Intensity Functional Training (HIFT)

SUMMARY:
Background Volleyball requires repeated explosive actions, agility, and technical precision, demanding contributions from both aerobic and anaerobic energy systems. Time-efficient training methods such as high-intensity interval training (HIIT) and high-intensity functional training (HIFT) have been proposed to enhance multidimensional performance in young athletes. However, direct comparisons of their effects in adolescent female volleyball players are limited.

Methods Thirty-two licensed female volleyball players (aged 15-18 years) were randomly assigned to HIIT (n=10), HIFT (n=11), or control (n=11). Training interventions lasted 12 weeks with two sessions per week, in addition to regular volleyball practice. The HIIT program consisted of progressive resistance-based high intensity intervals performed at 85-95% HRmax, while the HIFT program comprised multimodal circuit-style functional exercises performed at comparable intensities (~85-95% HRmax). Pre- and post-tests included countermovement jump (CMJ), standing long jump (SLJ), medicine ball throw (MBT), pro-agility, 20 m sprint, repeated sprint fatigue index (RSI), volleyball skill test, Yo-Yo IR1 distance, VO₂max, blood lactate, and maximal heart rate (MaxHR). A 3×2 mixed-model ANOVA with Tukey post hoc tests was conducted, and effect sizes were reported as Cohen's d and ηp².

DETAILED DESCRIPTION:
Volleyball is a high-intensity intermittent sport characterized by repeated explosive actions such as jumping, sprinting, accelerating, decelerating, and rapid changes of direction, combined with frequent technical maneuvers including serving, setting, spiking, and blocking. These actions require sustained neuromuscular output while maintaining technical precision under fatigue, placing substantial demands on both aerobic and anaerobic energy systems. Aerobic capacity is critical for sustaining recovery between rallies and maintaining performance throughout long matches or tournaments, whereas anaerobic power and strength are essential for explosive efforts that dominate competitive play. Additionally, agility, reactive strength, and coordination contribute significantly to performance, particularly in adolescent players who are still developing physiologically.

Given these demands, volleyball training requires conditioning approaches that are both time-efficient and sport-specific. Traditional continuous endurance training has been criticized for its poor transferability to volleyball, as it fails to replicate the intermittent, high-intensity, and multidirectional nature of the game. In contrast, modern approaches such as high-intensity interval training (HIIT) and high-intensity functional training (HIFT) have emerged as promising strategies. HIIT, involving repeated near-maximal bouts interspersed with structured recovery, has been shown to improve both aerobic and anaerobic capacity, enhance repeated sprint ability, and optimize recovery kinetics. However, resistance-based HIIT often emphasizes traditional strength exercises performed in a format with fixed rest intervals, which may not fully capture the sport-specific, multidirectional, and reactive movement patterns required in volleyball.

HIFT has been introduced as an integrative and multimodal training approach that combines plyometric drills, bodyweight resistance, agility exercises, and functional movements into circuit-based formats performed at high intensity with minimal recovery. Unlike resistance-based HIIT, which primarily involves structured strength exercises performed in a circuit format with fixed rest intervals, HIFT emphasizes more varied, compound, and task-oriented exercises that more closely mirror the sport-specific demands of volleyball. These exercises not only target cardiovascular fitness but also simultaneously improve explosive power, neuromuscular coordination, and stability. This integrative nature makes HIFT particularly promising for adolescent volleyball players, where physical conditioning must also support technical skill development and injury prevention.

Despite the growing use of both HIIT and HIFT in applied practice, direct experimental comparisons between these modalities in youth volleyball players are limited. Adolescence represents a critical developmental window where training adaptations can have long-term effects on physical performance, neuromuscular coordination, and resilience. Therefore, identifying the most effective training model for enhancing multidimensional performance in young female athletes is of high practical and scientific importance.

The present randomized controlled trial was designed to compare the effects of 12 weeks of HIIT and HIFT on performance outcomes in adolescent female volleyball players. Thirty-two licensed athletes aged 15-18 years, competing in a regional league, were randomly allocated into three groups: HIIT (n=10), HIFT (n=11), and a control group (n=11). All groups continued routine volleyball training (3-4 sessions per week). In addition, the intervention groups performed two supervised conditioning sessions weekly for 12 weeks, while the control group engaged in additional volleyball practice sessions to balance training volume.

Participants in the HIIT group engaged in a 12-week resistance-based high intensity interval training program, designed to target both aerobic and anaerobic energy systems. Training sessions were conducted twice per week in addition to the athletes' regular volleyball practice schedule. Each session commenced with a standardized 10-minute warm-up involving low-intensity jogging and dynamic stretching, and concluded with a 5-minute cool-down of light jogging and static stretching to promote recovery. The main training component consisted of short, repeated high intensity bouts (30 s) of multi-modal exercises-including sprint drills, plyometric movements, functional bodyweight resistance exercises, multi-joint strength movements, agility drills, and aerobic conditioning-performed at 85-95% of maximal heart rate (HRmax) Each bout was followed by 30 s of active recovery (e.g., walking or light movement).

Participants completed a 12-week high intensity functional training program aimed at developing aerobic capacity, anaerobic power, muscular strength, and agility. Training sessions were performed twice weekly in addition to regular volleyball practices. Each training session followed a standardized structure, beginning with a 10-minute warm-up of light jogging and dynamic mobility exercises, followed by a main training phase consisting of circuit-style functional workouts that combined sprint drills, plyometric exercises, bodyweight resistance movements, multi-joint strength exercises, agility drills, and aerobic activities; each exercise was performed for 30 seconds at maximal effort with no fixed rest between exercises (≤10 seconds transition allowed), and participants completed 4-6 sets per session with 1-2 minutes of rest between sets, while emphasizing maximal movement speed and explosive execution of all repetitions, and concluding with a 5-minute cool-down of low-intensity jogging and static stretching.

All performance assessments were conducted pre- and post-intervention under standardized laboratory and field conditions. The test battery included anthropometry and body composition, countermovement jump (CMJ), standing long jump (SLJ), medicine ball throw (MBT), pro-agility (5-10-5 shuttle run), 20 m sprint, repeated sprint fatigue index (RSA), volleyball skill test (serve, pass, set, block, spike), Yo-Yo Intermittent Recovery Test Level 1 (YYIR1), maximal oxygen uptake (VO₂max), blood lactate, maximal heart rate, and ratings of perceived exertion. Testing followed standardized warm-up and rest protocols, and measurements were conducted using validated equipment and procedures.

Ethical approval was obtained from the Marmara University Faculty of Medicine Clinical Research Ethics Committee (Protocol no: 09.2021.06; Date: January 8, 2021). Written informed consent was obtained from all participants and their legal guardians. COVID-19 regulations set by the Turkish Ministry of Health and the Ministry of Youth and Sports were strictly followed. Training and testing were supervised by qualified sport scientists and licensed coaches, with heart rate responses continuously monitored to ensure adherence to prescribed intensity zones.

ELIGIBILITY:
Inclusion Criteria:

* Female volleyball players aged 15-18 years
* Licensed athletes competing in a regional league
* Minimum of 2 years of regular volleyball training experience
* Healthy, without chronic illness or musculoskeletal injury
* Provided informed consent (with parental/guardian approval for minors)

Exclusion Criteria:

* Current musculoskeletal injury or recent surgery
* History of chronic disease (e.g., cardiovascular, metabolic, respiratory)
* Regular use of medication, nutritional supplements, alcohol, or tobacco
* Non-compliance with training sessions or inability to complete testing procedures
* Decline of informed consent or parental permission

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Countermovement Jump (CMJ) Height | Change from baseline to week 12
  Vertical jump height assessed using infrared timing device to evaluate explosive lower-limb power.
Change in Maximal Oxygen Uptake (VO₂max) | Change from baseline to week 12
  Measured using portable breath-by-breath metabolic analyzer during Yo-Yo IR1; reflects aerobic capacity.
Change in Volleyball Skill Test Score | Change from baseline to week 12
  Serve, pass, set, block, and spike accuracy under standardized conditions.

SECONDARY OUTCOMES:
Standing Long Jump (SLJ) Distance | Change from baseline to week 12
  Horizontal jump distance (cm) to assess lower-limb power.
Medicine Ball Throw Distance | Change from baseline to week 12
  Seated chest-pass with 3-kg medicine ball to assess upper-limb explosive strength.
Pro-Agility Test (5-10-5 Shuttle) | Change from baseline to week 12
  Change-of-direction speed measured with electronic timing gates (s).
20 m Sprint Time | Change from baseline to week 12
  Linear sprint performance measured in seconds.
Repeated Sprint Fatigue Index (RSI) | Change from baseline to week 12
  Percentage decline across 10 × 20 m sprints.
Yo-Yo Intermittent Recovery Test Level 1 Distance | Change from baseline to week 12
  Total distance covered (m) to assess intermittent aerobic endurance.
Blood Lactate Concentration | Change from baseline to week 12
  Capillary blood lactate (mmol/L) pre- and post-YYIR1.
Maximal Heart Rate (MaxHR) | Change from baseline to week 12
  Peak heart rate (bpm) during YYIR1.
Rating of Perceived Exertion (RPE) | Change from baseline to week 12
  Perceived exertion was assessed using the Borg Rating of Perceived Exertion Scale (6-20 points) immediately following the Yo-Yo Intermittent Recovery Test Level 1 (YYIR1).
  On this scale, 6 indicates "no exertion at all" and 20 indicates "maximal exertion." Higher scores represent a greater level of perceived exertion (i.e., a worse outcome in terms of subjective fatigue).

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Faculty of Sport Sciences Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional and ethical restrictions

REFERENCES:
- [Derived] Bilici OF, Topates TK. Comparative effects of high intensity interval and functional training on performance outcomes in adolescent female volleyball players. BMC Sports Sci Med Rehabil. 2025 Dec 23. doi: 10.1186/s13102-025-01476-w. Online ahead of print. PMID 41437127